CLINICAL TRIAL: NCT04083677
Title: Lecturer of Anesthesia
Brief Title: Routine Point of Care Ultrasound (POCUS) Assessment of Antral Gastric Contents in Traumatic Surgical Patients for Prevention of Aspiration Pneumonitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, lecturer of anesthesia at faculty of medicine ain shams university, Ain Shams University
Other Study IDs: Ain Shams university 11
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control GROUP: healthy adult fasting 8 hours before the operation sonographic examination of gastric antrum before anesthesia
  Interventions: Device: SONAR
- trauma GROUP: trauma patients fasting 8 hours before the operation sonographic examination of gastric antrum before anesthesia
  Interventions: Device: SONAR

INTERVENTIONS:
Device: SONAR — A curved low- frequency (2-5 MHZ) probe and (simens ACUSON x 300) ultrasound system will be used. All patient will be first scanned in the supine position, followed by the right lateral decubitus (RLD) position. The gastric antrum was identified in a sagittal scanning plane in the epigastrium immediately inferior to xiphoid and superior to umbilicus. The liver anteriorly and the aorta, inferior vena cava and pancreas posteriorly were used as anatomical reference points.

SUMMARY:
Pulmonary aspiration of gastric contents is uncommon in the elective, surgical populations, but highly prevalent in trauma patients who requires emergency surgery as trauma impair gastric motility and emptying.1 Presence of residual gastric volume at the time of anesthetic induction is an important risk of aspiration pneumonitis.2 Routine use of non-invasive bedside ultrasound gives information about the volume and nature of gastric volume. Determination of gastric content volume preoperatively will help the anesthetist in the assessment of pulmonary aspiration risk 3, 4 Ultrasongraphic measurment of antral CSA (cross sectional area) can diagnose risk stomach during the preoperative period defined by a gastric volume at risk of pulmonary aspiration (ie presence of Solid particles and/or gastric volume >1.5 ml/kg)5 The aim of our study is to allow routine use of point of care ultrasound (pocus) of gastric contents in order to inform an assessment of aspiration risk and guide anesthetic mangment

DETAILED DESCRIPTION:
A prospective randomized study will be conducted in Ain Shams University Hospital-Emergency Department. Institutional Research Ethics Committee approval will be obtained and written informed consent will be obtained from all participants before enrollment. The study included forty five polytrauma patients (18-65 years old of both sexes) admitted for emergency surgery.

On admission, ABC protocol will be applied, (GCS) Glasgow coma scale assessment, complete laboratory investigations and radiology and complete clinical examination with assessment of fasting hours.

Exclusion criteria are patients with obesity (BMI> 35kg/m2), pregnancy, a history of upper gastrointestinal diseases including gastroesophageal reflux disease, hiatus hernia, gastroeosphgeal cancer or upper GIT surgery.

A curved low- frequency (2-5 MHZ) probe and (simens ACUSON x 300) ultrasound system will be used. All patient will be first scanned in the supine position, followed by the right lateral decubitus (RLD) position. The gastric antrum was identified in a sagittal scanning plane in the epigastrium immediately inferior to xiphoid and superior to umbilicus. The liver anteriorly and the aorta, inferior vena cava and pancreas posteriorly were used as anatomical reference points.

Fig. (1): Sagittal/parasgittal scanning plane for gastric assessment

Fig. (2) A Sagittal sonogram of the gastric antrum. A = antrum; L = liver; P = pancreas; SMA = superior mesenteric artery; Ao = aorta. B Schematic representation of sagittal sonoanatomy. A = antrum; L = liver; P = pancreas; SMA = superior mesenteric artery; Ao = aorta

The "empty" antrum appeared collapsed and "flat" with the anterior and posterior walls very close to each other or round to ovoid in shape resembling a "bull's eye" target.

The antrum appeared distended with a round shape when filled with a clear fluid. Multiple gas "bubbles" appeared as punctuate hyperechoic areas within the hypoechoic fluid, mimicking a "starry night" appearance.

The antrum appeared distended with a contents of mixed echogenicity when filled with a solid contents give the antrum "frosted glass" appearance.

When the stomach contains clear fluid, a volume assessment can help differentiate a negligible volume consistent with baseline secretions vs a higher than baseline volume. So, the antral cross sectional area (CSA) was calculated after measuring the two dimensions of the antrum (D1 an D2) according to the following equation: π (D1 x D2)/4 and the volume of clear fluid was calculated using a cross- sectional area CSA of the antrum measured in the RLD and a previously published mathematical model: volume (ml)= 27.0+(14.3 x Right - lat (CSA) - (1.25 x age). This equation accurately predicts gastric volume up to 500 ml.

Nasogastric ryle will be inserted (if there is no contraindication) to confirm gastric ultrasound volume calculation.

Additionally, the antrum as classified according to a 3-point grading system (perlas grade 0-2) that is based on the absence or presence of clear fluid in the supine and RLD positions. Grade 0 refers to the absence of gastric content in the antrum in both supine and RLD positions. Grade 1 refers to antral clear fluid that is appreciable only in the RLD. Grade 2 refers to clear fluid that is documented in both the supine and RLD positions.

Fig.(3): flow chart for interpretation of findings and medical decision- making based on gastric point of care ultrasound findings. Used with permission from gastric ultrasound. Org The low risk result will suggest that the risk of aspiration is low and it may be safe to proceed with surgery with a slowly titrated induction of anesthesia as dictated by the patient's cardiac condition using laryngeal mask or E.T.T.

The high risk result will suggest that the risk of aspiration is high, and this finding would support: 1, postponing surgrery, till completion of fasting hours 2 loco-regional anesthesia; neuraxial anesthesia, and 3, general anesthesia with rapid sequence induction, up to awake fibro-optic intubation.

We will record the incidence of change in anesthetic technique and change in timing of surgical procedure (as a primary outcome) and incidence of perioperative aspiration (as a secondary outcome) when we use gastric ultrasound preoperatively in these patients.

Sample size:

Using medical program setting alpha error at 5% & power at 90% we calculated our sample size based on the result of (sabry et al., 2018) which showed very good correlation between gastric volume using ultrasound and volume of aspirated gastric content with an assumed (r=0.5). Based on this the needed sample is 45 cases taken in account 10% drop out rate.

ELIGIBILITY:
Inclusion Criteria:

* polytrauma patients admitted for emergency surgery.

Exclusion Criteria:

* patients with obesity (BMI> 35kg/m2),
* pregnancy,
* a history of upper gastrointestinal diseases including gastroesophageal reflux disease, hiatus hernia, gastroeosphgeal cancer or upper GIT surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included forty five polytrauma patients (18-65 years old of both sexes) admitted for emergency surgery.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
gastric content | 6 months
  gastric content volume by sonar

CONTACTS AND LOCATIONS:
Overall Officials: ramy mahrose, md, Study Director — asuh
Locations (1):
- Ramymahrose, Cairo, Egypt

REFERENCES:
- [Derived] Shorbagy MS, Kasem AA, Gamal Eldin AA, Mahrose R. Routine point-of-care ultrasound (POCUS) assessment of gastric antral content in traumatic emergency surgical patients for prevention of aspiration pneumonitis: an observational clinical trial. BMC Anesthesiol. 2021 May 8;21(1):140. doi: 10.1186/s12871-021-01357-y. PMID 33964867 (Retraction: PMID 35864458 BMC Anesthesiol. 2022 Jul 21;22(1):233)